CLINICAL TRIAL: NCT06944418
Title: The Study of Differences in Eosinophil Function and Subsets in Patients With Eosinophilic Pulmonary Diseases Based on Flow Cytometry Analysis
Brief Title: The Study of Differences in Eosinophil Function and Subsets in Patients With Eosinophilic Pulmonary Diseases
Status: Recruiting | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-EPD
Record Dates: First submitted 2025-03-30; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Eosinophil Subtype; Eosinophilic Pulmonary Diseases
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: observation — observation

SUMMARY:
The study subjects of this research are patients with eosinophil-associated pulmonary diseases, including eosinophilic granulomatosis with polyangiitis, idiopathic hypereosinophilic syndrome, idiopathic acute eosinophilic pneumonia, idiopathic chronic eosinophilic pneumonia, and primary simple pulmonary eosinophilia. The aim is to detect eosinophil subtypes in peripheral blood based on surface protein expression, to understand the differences in eosinophil subtypes among patients with different diseases, to elucidate the significance of different eosinophil subtypes, and ultimately to provide a theoretical basis for the selection of treatment directions for patients.

ELIGIBILITY:
Inclusion Criteria:

* For Healthy Volunteers: healthy volunteers matching the age and gender of the study subjects
* For EPD: ① Persistent eosinophil count increase>1500 per cubic millimeter for more than 6 months. ② Lack of evidence of a secondary cause of eosinophilia is required. ③ Signs and symptoms of end-organ damage presumed to be secondary to eosinophilia

Exclusion Criteria:

* Patients with concurrent definitive pulmonary infections, malignancies, or other parenchymal lung diseases;
* Patients who are unable or unwilling to cooperate with the collection of clinical information (e.g., due to mental disorders, memory impairments, etc.);
* Patients who are unable to provide informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Outpatients diagnosed with EPD who meet the inclusion criteria above.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of Eosinophil Subtypes in Serum | From January 1, 2024 to January 1, 2027
  Proportion of Eosinophil Subtypes in Serum Before and After Treatment in Patients

CONTACTS AND LOCATIONS:
Overall Officials: Juhong Shi, M.D, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No